CLINICAL TRIAL: NCT04951544
Title: Pilot-test of an mHealth Black Men Who Have Sex With Men (MSM) in Couples Intervention (LetSync v1.0, v2.0)
Brief Title: LetSync: Pilot Test of Mobile Health (mHealth) Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 5R01MH118967-03 (NIH); 5R01MH118967-03 (NIH)
Record Dates: First submitted 2021-06-16; First posted 2021-07-07 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: HIV/AIDS
Keywords: HIV/AIDS; mHealth; Intervention; African American men
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): This arm will start the intervention using LetSync app v1.0 from T1 to T4, baseline/Month 0 to Month 14.
  Interventions: Other: LetSync v1.0
- Waitlist-Control Group (Active Comparator): This arm will wait to begin the intervention using the LetSync app v2.0 from T3 to T4, Month 8 to Month 14.
  Interventions: Other: LetSync v2.0

INTERVENTIONS:
Other: LetSync v1.0 — Study B will entail a pilot randomized, controlled trial (RCT) of an mHealth behavioral intervention, LetSync, with 80 couples (N=160) to assess its acceptability, feasibility, and preliminary impact on retention in care and ART adherence as measured by antiretroviral concentrations in hair. Participants in the intervention arm will use LetSync v1.0 for 6 months and provide acceptability and feasibility data. Participants will then continue to use LetSync v1.0 while the Waitlist-Control group begins to use LetSync v2.0.
  Arms: Intervention Group
Other: LetSync v2.0 — LetSync v2.0 will be developed by taking feedback from participants regarding LetSync v1.0. Participants in the waitlist-control group will be given LetSync v2.0 to use during the last 6 months of the trial.
  Arms: Waitlist-Control Group

SUMMARY:
The Pilot Test (AKA Study B) will entail a pilot randomized, controlled trial (RCT) of an mHealth behavioral intervention, LetSync, with 80 couples (N=160) to assess its acceptability, feasibility, and preliminary impact on retention in care and ART adherence as measured by antiretroviral concentrations in hair. Participants in the intervention arm will use LetSync v1.0 for 6 months and provide acceptability and feasibility data. In the ensuing 2 months, the investigators will make refinements based on participants' data to produce LetSync v2.0. Then, participants in the waitlist-control arm will receive LetSync v2.0, use it for 6 months, and provide acceptability and feasibility data. The intervention arm will continue using LetSync v1.0, for a total of 14 months. Based on acceptability and feasibility data from waitlist control arm participants between T3 and T4, the investigators will develop LetSync v3.0, which will be used for efficacy testing in a full RCT trial in the future.

ELIGIBILITY:
Inclusion Criteria:

Individuals are eligible if they:

* Self-identify as racial/ethnic minority
* Self-identify as a cisgender man
* Are HIV-Positive themselves, or are the partner of someone who is living with HIV
* Are age 18 or older
* Have a primary relationship partner, defined as someone to whom the participant is committed above anyone else for three or more months
* Uses and owns a personal smartphone
* Willing and able to provide informed consent

Partners are eligible if they:

* Self-identify as a cisgender man
* Are age 18 or older
* Have a primary relationship partner that is the referring participant
* Uses and owns a personal smartphone
* Willing and able to provide informed consent

Exclusion Criteria:

Those who:

* Report fear of intimate partner violence (IPV) resulting from participation
* Are unwilling or unable to disclose HIV status to primary partner
* Present evidence of severe cognitive impairment that would prevent comprehension of study procedures assessed during informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must identify as a cis-gender man - that is, they must currently identify as a man and have been born a male.
Enrollment: 144 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Levels of Antiretroviral (ARV) concentration in dried blood spot (DBS) samples | 8 months
  The investigators will use the UNC Pharmacology Lab to analyze ARV levels in dried blood spot (DBS) samples as an objective measure of drug adherence and exposure for HIV-infected participants. The investigators will mail participants a DBS sample collection kit with necessary supplies, detailed instructions via online demonstration video, and a prepaid return envelope. DBS samples will be collected and analyzed between baseline (T0) and 8 months (T4).
  ARV levels will be measured as nanograms per milligram (ng/mg) of DBS will be log-transformed for data analysis. Changes since Baseline of ARV levels will be measured.
Self-reported measure of care engagement | 8 months
  Self-reported care engagement will be measured with the 10-item Index of Engagement in HIV Care rated on a Likert-type scale ranging from 1 to 5, 'Strongly disagree' to 'Strongly agree'. This will be included in questionnaires administered to participants between baseline (T0) and 8 months (T4).
  A mean Index score will be calculated (the sum of all items without missing responses divided by that number of items), with a higher score representing better care engagement and lower score representing worse care engagement. Changes since Baseline of the mean Index score will be measured.
Self-reported measure I of antiretroviral therapy (ART) adherence | 8 months
  Self-reported antiretroviral therapy (ART) adherence will be measured using an aggregated or composite score derived from the following items. Frequency of missed doses will be represented by summing the following two items: how many doses were missed over the last 30 days, and how many doses missed over the past three months for at least four days in a row.
Self-reported measure II of antiretroviral therapy (ART) adherence | 8 months
  Self-reported antiretroviral therapy (ART) adherence will be measured using an aggregated or composite score derived from the following items on a Likert-type scale of 1 to 5, 'Strongly disagree' to 'Strongly agree': Self-rated ability of taking medications the way they should, how often they took medications the way they should.
  For self-rated ability of taking medications and frequency of taking them, a mean score will be calculated (the sum of all items without missing responses divided by that number of items). A higher score represents excellent ability of taking medications and a lower score represents poor ability of taking medications. Changes in Baseline for the mean Index score will be measured.
Presence of Antiretroviral (ARV) medication in urine sample | 8 months
  The investigators will use self-collected urine samples as another objective measure of drug adherence for participants living with HIV. The investigators will mail participants a urine sample collection kit with necessary supplies and detailed instructions via online demonstration video. Participants will self-collect and administer the urine sample and send a photo of the results to study staff. Urine test results will be collected between baseline (T0) and 8 months (T4).

SECONDARY OUTCOMES:
Feasibility or usability of LetSync app v1.0 (how easy or convenient is v1.0 to use) | 8 months
  Between baseline (T0) and 8 months (T4), the investigators will collect feasibility-related data via the app using a validated 10-item Feasibility instrument. The items are on a five-point Likert scale ranging from 'Strongly disagree' to 'Strongly agree'. A mean Feasibility score will be calculated (the sum of all items without missing responses divided by that number of items). A higher score indicates high feasibility, whereas a lower score indicates low feasibility.
  Feasibility data collected only between baseline (T1) and 6 months (T2) will be used to develop LetSync app v2.0 for the Waitlist-control arm. Investigators will continue collecting acceptability data on LetSync app v1.0 from the Intervention arm.
Acceptability of or Satisfaction in using LetSync app v1.0 | 8 months
  Between baseline (T0) and 14 months (T5), the investigators will collect acceptability data via the app using a validated 5-item Feasibility instrument. The items are on a five-point Likert scale (1 to 5) ranging from 'Strongly disagree' to 'Strongly agree'. A mean Acceptability score will be calculated (the sum of all items without missing responses divided by that number of items). A higher score indicates high acceptability, whereas a lower score indicates low feasibility.
  Acceptability data collected only between baseline (T1) and 6 months (T2) will be used to develop LetSync app v2.0 for the Waitlist-control arm. Investigators will continue collecting acceptability data on LetSync app v1.0 from the Intervention arm.
Self-reported care engagement | 8 months
  The investigators will collect data on participants' self-reported care engagement; this will be comprised of scheduled, cancelled, rescheduled, and attended visits to their HIV and/or primary care provider within the last three to six months. Data will be collected via questionnaires administered to participants between baseline (T0) and 8 months (T4). The investigators will measure changes from Baseline for each item of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Judy Y Tan, Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim HC, Pollack LM, Saberi P, Neilands TB, Arnold EA, Bright DJ, Williams RW, Kegeles SM, Tan JY. Study protocol: a pilot randomised waitlist-controlled trial of a dyadic mobile health intervention for black sexual-minority male couples with HIV in the USA. BMJ Open. 2021 Sep 2;11(9):e055448. doi: 10.1136/bmjopen-2021-055448. PMID 34475191